CLINICAL TRIAL: NCT05566756
Title: A Non-interventional Study Evaluating Kesimpta® (Ofatumumab) Treatment Effects in Patients With Relapsing Multiple Sclerosis Transitioning From Other Therapies [KAIROS]
Brief Title: Study Evaluating Kesimpta® Treatment Effects in Patients With Relapsing Multiple Sclerosis Transitioning From Other Therapies
Acronym: KAIROS
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GDE03
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; MS; Kesimpta; ofatumumab
MeSH Terms: conditions — Multiple Sclerosis | interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ofatumumab: Patients prescribed with ofatumumab
  Interventions: Other: Ofatumumab

INTERVENTIONS:
Other: Ofatumumab — There is no treatment allocation. Patients administered Ofatumumab by prescription will be enrolled.
  Other Names: Kesimpta

SUMMARY:
KAIROS is a prospective, multicenter, non-interventional study (NIS) in Germany. Prospective, primary data will be collected via questionnaires and an electronic case report form (eCRF) over a period of one year (max. 1.5 years) of treatment. Additionally, medical history of participants will be collected including disease duration, EDSS, MRI parameters and relapses.

DETAILED DESCRIPTION:
The decision for ofatumumab as routine medical treatment must be taken independently of and prior to the study start. During the observation phase of the study, data will be collected according to standard of care as recommended by KKNMS (Competence Network Multiple Sclerosis in Germany).

The prospective observational period per patient will be up to approx. one year from the time of consent (1 year ± 2 months visit window + potentially 6 months follow-up to confirm disability worsening in patients who showed increase in EDSS within 6 months prior to EOS). The observational period will not be dictated by the protocol. The follow-up documentation will take place at a frequency defined as per investigator's discretion. The diagnostic or monitoring procedures are only those ordinarily applied to the therapeutic strategy and to routine clinical care, can be performed as telemedicine visits and will take place as per investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before participating in the study
2. Diagnosis of RMS per McDonald Criteria (2017) (Thompson, Banwell et al. 2018)
3. Prior treatment with EU approved DMT for MS other than ofatumumab
4. Decision for treatment initiation of ofatumumab (Kesimpta®) prior to study participation and planned initiation of ofatumumab after respective wash-out period of prior DMT (if applicable) or performed initiation of ofatumumab within the last 14 days
5. Ofatumumab treatment in line with the German label

Exclusion Criteria:

1. Use of investigational drugs during the study, OR within 3 months before ofatumumab initiation, OR within 5 half-lives of investigational drug before ofatumumab initiation, OR until the expected pharmacodynamic effect has returned to baseline, whichever is longer
2. Subjects who are not able to provide consent due to incapable judgement
3. Simultaneous participation in any investigational trial or simultaneous participation in another Novartis-sponsored non-interventional study with ofatumumab

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who previously received any approved DMT for RMS in Germany, and the decision to transition to ofatumumab therapy due to safety, tolerability, efficacy or other reasons was taken, will be eligible for enrollment
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Reasons for recent therapy switch to ofatumumab | Baseline
  Reasons for recent therapy switch to ofatumumab will be collected

SECONDARY OUTCOMES:
Proportion of missed ofatumumab doses | 12 months
  Proportion of missed ofatumumab doses within one year, defined as the difference between number of planned doses and number of administered doses
Number of patients by reasons for treatment interruptions | 12 months
  Reasons for treatment interruptions per patient will be collected
Number of treatment interruptions per patient | 12 months
  Number of treatment interruptions per patient will be collected
Duration of treatment interruptions per patient | 12 months
  Duration of treatment interruptions per patient will be collected
Proportion of patient subgroups with and without 100% adherence depending on different characteristics | 12 months
  Proportion of patient subgroups with and without 100% adherence depending on different characteristics, defined as patients with matching number of planned doses and number of administered doses within 1 year (e.g., previous experience with sub-cutaneous therapy)
Proportion of patients permanently discontinuing ofatumumab during the study by reason for discontinuation | 12 months
  Proportion of patients permanently discontinuing ofatumumab during the study by reasons for discontinuation will be collected
Proportion of patients permanently discontinuing ofatumumab during the study by planned next DMT | 12 months
  Proportion of patients permanently discontinuing ofatumumab during the study by planned next DMT
Change on Multiple Sclerosis Impact Scale 29 (MSIS-29) as compared to baseline in general and depending on reasons for treatment switch | Baseline, month 6, month 12
  MSIS-29 is a 29-item, self administered questionnaire that includes two domains, physical and psychological. Responses are captured on a 4-point scale ranging from "not at all" (1) to "extremely" (4), where higher scores reflect greater impact on day-to-day life.
  The questions in the scale ask the subjects for their views about the impact of MS on their day to-day life during the past 2 weeks.
  Analysis will be done depending on the reasons for treatment switch.
Treatment Satisfaction Questionnaire for Medication (TSQM) 1.4 as compared to baseline in general and depending on reasons for treatment switch | Baseline, month 6, month 12
  The TSQM Version 1.4 comprises 14 items across four domains focusing on effectiveness (3 items), side effects (5 items), convenience (3 items), and global satisfaction (3 items) of the medication over the previous 2-3 weeks, or since the subject´s last use. With the exception of item 4 (presence of side effects; yes or no), all items have 5 or 7 responses, scored from 1 (least satisfied) to 5 or 7 (most satisfied). 7-item scales had a non-neutral midpoint, such that there were more positive response options than negative response options, to allow precise information to be obtained at the upper end of the score distribution. Item scores are summarized to give four domain scores, which are in turn transformed to a scale of 0
  -100.
Fatigue Scale for Motor and Cognitive Functions (FSMC) compared to baseline in general and depending on reasons for treatment switch | Baseline, month 6, month 12
  FSMC is a 20 item scale developed as a measure of cognitive and motor fatigue for people with Multiple Sclerosis.
  Each item is rated on a scale from 1-5 (1:"does not apply", 5: "applies completely").
  Thus, a maximum of 100 points for the total scale can be achieved. A patient who has neither motor nor cognitive fatigue would thus achieve a score of 20 for the total scale.
Percentage of patients with no clinical evidence of disease activity (NEDA) | Baseline, month 6, month 12
  NEDA is defined by no confirmed MS relapse, no new or enlarging T2 lesions, no Gadolinium-positive T1 lesions, and no six-month confirmed disability worsening
Proportion of patients demonstrating the individual NEDA-3 components | Baseline, month 12
  The individual NEDA-3 components are:
  * proportion of patients with no confirmed MS relapse
  * proportion of patients with no new or enlarging T2 lesions and no Gadolinium-positive T1 lesions
  * proportion of patients with no six-month confirmed disability worsening
The proportion of subjects discontinuing treatment due to insufficient effectiveness (lack of effectiveness) or tolerability/safety reasons | 12 months
  The proportion of subjects discontinuing treatment due to insufficient effectiveness or tolerability/safety reasons
Number of participants with injection related AEs | 12 months
  injection site reaction AEs vs. injection systemic reaction AEs

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- Germany (35):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Bamberg, Bavaria
  - Novartis Investigative Site, Bad Homburg, Hesse
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Altenburg, Thuringia
  - Novartis Investigative Site, Alzey
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bogen
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Gelsenkirchen
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Gladenbach
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kaiserslautern
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Pforzheim
  - Novartis Investigative Site, Quakenbrück
  - Novartis Investigative Site, Remscheid
  - Novartis Investigative Site, Rülzheim
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Sinsheim
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Unterhaching

IPD SHARING:
Plan to Share IPD: No